CLINICAL TRIAL: NCT03353922
Title: Driving Simulation Cross-Over Study of Sedative Effects of Tolperisone Compared to Cyclobenzaprine and Placebo
Brief Title: Driving Simulation to Assess Non-Sedative Effects of Tolperisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurana Pharmaceuticals, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NR115
Record Dates: First submitted 2017-11-14; First posted 2017-11-27 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Driving Impaired
Keywords: cognitive function
MeSH Terms: interventions — cyclobenzaprine; Tablets

STUDY DESIGN:
Intervention Model Description: multiple-dose 3-way cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: subjects are blindfolded to receive oral dose of treatment, matching placebo, or unblinded active control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tolperisone HCl 150 mg (Experimental): 150 mg tolperisone tablets or cyclobenzaprine 10 mg oral tablet administered by mouth every 8 hours for 3 days
  Interventions: Drug: Cyclobenzaprine 10 Mg Oral Tablet; Drug: Placebo Oral Tablet
- Placebo Oral Tablet (Placebo Comparator): sugar pills administered by mouth every 8 hours for 3 days
  Interventions: Drug: Cyclobenzaprine 10 Mg Oral Tablet; Drug: Placebo Oral Tablet
- Cyclobenzaprine 10 mg oral tablet (Active Comparator): 10 mg cyclobenzapine tablets administered by mouth every 8 hours for 3 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Cyclobenzaprine 10 Mg Oral Tablet — cyclobenzaprine 10 mg tablets
  Other Names: Flexeril
  Arms: Placebo Oral Tablet; Tolperisone HCl 150 mg
Drug: Placebo Oral Tablet — sugar pill
  Other Names: tolperisone matching placebo

SUMMARY:
This is a randomized blinded study to assess the sedative effect of 150 mg TID tolperisone and 10 mg TID cyclobenzaprine compared to placebo on simulated driving performance and cognitive functioning in healthy adult volunteers.

DETAILED DESCRIPTION:
This will be a randomized, placebo-controlled, multiple-dose 3-way cross-over study of the safety and cognitive effects of multiple doses of 150 mg tolperisone administered TID in 30 male and female healthy volunteers. Treatment groups include 450 mg tolperisone (i.e., 150 mg administered three times daily), 30 mg cyclobenzaprine (i.e., 10 mg administered three times daily), and placebo. Subjects will receive 3 days of each treatment.

Subject participation will be approximately 3 weeks as outpatients with 3 days each week as overnight clinic participants.

In this crossover study, treatment effects will be assessed following the second initial dose, the morning following nighttime dosing (to assess residual next day effects), and at steady state (i.e., following AM dosing on Day 3).

Subjects will be dosed on the morning of Day 1. Approximately one hour after the second dose on Day 1, subjects will be administered the cognitive test, followed by the driving simulator examination.

On the morning of Day 2, prior to dosing, subjects will be readministered the cognitive test and driving examination to assess residual next day effects.

Subjects will repeat cognitive testing and the driving examination on the morning of Day 3, after administration of the AM study medication, to evaluate the cumulative effects of 3 days of dosing.

ELIGIBILITY:
Inclusion Criteria:

1. All healthy volunteer subjects must be in general good health based on screening physical examination (defined as the absence of any clinically relevant abnormalities), medical history, 12-lead ECG, and clinical laboratory values (hematology, serum chemistry and urinalysis).
2. All subjects must be capable of understanding and complying with the protocol and have signed the informed consent document. Female subjects of childbearing potential must sign the Women of Childbearing Potential Addendum to the informed consent form.
3. Subjects are required to have a body mass index (BMI) of 18 to 32 kg/m2, inclusive, at Screening.
4. Subject must be able to reliably perform study assessments (i.e., SDLP no higher than 1 standard deviation greater than the mean for normal healthy adults completing the CVDA practice scenario; and number correct on CogScreen Symbol Digit Coding no less than 1 standard deviation below the mean for healthy adults in the 21-55 year age range); demonstrates the ability to understand task instructions (in English), and be physically capable (e.g., adequate manual dexterity, vision, and hearing), cognitively capable and motivated to perform study tasks.
5. Subject must possess a valid driver's license and be an active driver, and have driven a minimum of 10,000 miles (about 16,000 km) per year for the previous 3 years.
6. Subject must also demonstrate simulator sickness questionnaire scores which are not indicative of simulator sickness as defined in the driving simulation operations manual.
7. Subject must have a regular sleep pattern, not be engaged in shift-work, and in general, have at least 7 hours of sleep each night (bedtime occurs between 21:00 and 24:00 hours).
8. Subject has a score < 10 on the Epworth Sleepiness Scale (ESS).
9. Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Subjects who have any clinically significant unstable medical abnormality, chronic disease or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems.
2. Subjects who test positive at screening for hepatitis B surface antigen, hepatitis C antibody or have a history of a positive result.
3. Subjects who are known to be seropositive or test positive at Screening for Human immunodeficiency virus (HIV).
4. Female subjects who are pregnant or lactating.
5. Subjects who have a disorder or history of a condition (e.g., malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
6. A history within 2 years of, or current treatment for a sleeping disorder (including excessive snoring, obstructive sleep apnea), or a chronic painful condition that interferes with the subject's sleep.
7. A history of difficulty in falling asleep or staying asleep in the previous 3 months, that is considered clinically significant by the investigator.
8. Subjects who have a history or diagnosis of any of the following conditions:

   1. Primary or secondary insomnia
   2. Narcolepsy
   3. Cataplexy (familial or idiopathic)
   4. Circadian Rhythm Sleep Disorder
   5. Parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and rapid eye movement behavior disorder
   6. Sleep-related Breathing Disorder (obstructive or central sleep apnea syndrome, central alveolar hypoventilation syndrome)
   7. Periodic Limb Movement Disorder
   8. Restless Legs Syndrome
   9. Primary Hypersomnia
   10. Excessive Daytime Sleepiness (EDS)
   11. Subject has visual or auditory impairment which in the opinion of the investigator would interfere with study related procedures or study conduct.
9. Subjects expected to use any other medication or dietary supplement to promote sleep including over-the-counter sleep medications, during their participation in the study.
10. Subjects who have participated in any investigational study within 30 days prior to screening or are currently participating in another clinical trial.
11. Subjects who have had a recent history (less than 2 years before entering the study) of drug or alcohol abuse, or current positive urine drug screen. Alcohol abuse is defined as current consumption of more than three alcoholic beverages per day.
12. Subjects who have a history of allergic reaction to tolperisone or cyclobenzaprine or any components of these study medications.
13. Use of psychoactive prescription or non-prescription medications, psychoactive nutritional supplements or herbal preparations within 2 weeks or 5 half-lives (whichever is longer) of admission to the Clinical Research Unit (CRU) on Day 1.
14. Presence of a medical or psychiatric condition which could jeopardize the safety of the subject or validity of study results
15. Subjects who consume excessive amounts of coffee, tea, cola, or other caffeinated beverages per day. Excessive amount is defined as greater than 6 servings per day (where 1 serving is approximately equivalent to 120 mg of caffeine).
16. Subjects who will be working a night shift within 1 week of a visit.
17. Subject who have traveled across 1 or more time zones (transmeridian travel) in the last 2 weeks prior to randomization or is expected to travel across 1 or more time zones during the study.
18. Current smoker (>10 cigarettes or eCigarettes, 3 cigars, or 3 pipes per day) and unwilling to refrain from smoking while confined to the CRU for periods of 3 days.
19. Subjects who have an inability or unwillingness to abide by the study protocol or cooperate fully with the Investigator or designee.
20. Subjects who are a staff member or relative of a staff member.
21. Inability or unwillingness to use adequate contraception (as defined in item 10 of the Inclusion Criteria) during and for 1 month following completion of the study.
22. Has a positive screen for alcohol or other drugs of abuse (amphetamines, methamphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, Long Beach, California
  - NeuroTrials Research, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized 3-way cross-over of multiple doses of 150 mg tolperisone, 10 mg cyclobenzaprine, or placebo TID in 35 male & female healthy volunteers. Treatment groups A (Tolperisone), B (Cyclobenzaprine), and C (Placebo) randomized by 6 treatment sequences. Subjects serve as own positive control, data analyzed and reported based on treatment type.
Groups:
- ABC (Tolperisone, Cyclobenzaprine, Placebo): 1st intervention: 150 mg tolperisone tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: 10 mg cyclobenzaprine every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: placebo every 8 hours for 3 days, followed by release from clinic.
- ACB (Tolperisone, Placebo, Cyclobenzaprine): 1st intervention: 150 mg tolperisone tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: placebo every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: 10 mg cyclobenzaprine every 8 hours for 3 days, followed by release from clinic.
- BAC (Cyclobenzaprine, Tolperisone, Placebo): 1st intervention: 10 mg cyclobenzaprine tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: 150 mg tolperisone cyclobenzaprine every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: placebo every 8 hours for 3 days, followed by release from clinic.
- BCA (Cyclobenzaprine, Placebo, Tolperisone): 1st intervention: 10 mg cyclobenzaprine tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: placebo every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: 150 mg tolperisone every 8 hours for 3 days, followed by release from clinic.
- CAB (Placebo, Tolperisone, Cyclobenzaprine): 1st intervention: placebo tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: 150 mg tolperisone every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: 10 mg cyclobenzaprine every 8 hours for 3 days, followed by release from clinic.
- CBA (Placebo, Cyclobenzaprine, Tolperisone): 1st intervention: placebo tablets administered every 8 hours for 3 days, followed by washout period of 4 days, then 2nd intervention: 10 mg cyclobenzaprine every 8 hours for 3 days, followed by 4 day washout, then 3rd intervention: 150 mg tolperisone every 8 hours for 3 days, followed by release from clinic.
Period: Overall Study
Arm/Group | ABC (Tolperisone, Cyclobenzaprine, Placebo) | ACB (Tolperisone, Placebo, Cyclobenzaprine) | BAC (Cyclobenzaprine, Tolperisone, Placebo) | BCA (Cyclobenzaprine, Placebo, Tolperisone) | CAB (Placebo, Tolperisone, Cyclobenzaprine) | CBA (Placebo, Cyclobenzaprine, Tolperisone)
Started | 6 | 6 | 6 | 6 | 5 | 6
Completed (35 subjects signed consent; 4 discont.-3 withdrew consent before tx, 1 for AE in tolperisone tx arm) | 5 | 5 | 5 | 5 | 5 | 6
Not Completed | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Final analysis on per protocol population (n=33) instead of ITT (n=35) due to 2 subjects being mis-dosed
Groups:
- All Study Participants: All Study Participants; n=33
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants] — Population: Final analysis on per protocol population (n=33) instead of ITT (n=35) due to 2 subjects being mis-dosed
  Participants
    <=18 years | 0
    Between 18 and 65 years | 33
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Cross over design for subjects, not independent groups
  Participants
    Female | 10
    Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Final analysis on per protocol population (n=33) instead of ITT (n=35) due to 2 subjects being mis-dosed
  Participants
    Hispanic or Latino | 10
    Not Hispanic or Latino | 23
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Final analysis on per protocol population (n=33) instead of ITT (n=35) due to 2 subjects being mis-dosed
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 15
    White | 17
    More than one race | 0
    Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m2] — kg/m2 Population: Final analysis on per protocol population (n=33) instead of ITT (n=35) due to 2 subjects being mis-dosed
  kg/m2 | 25.012 (2.959)

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation of Lateral Position (SDLP)
Description: In this crossover study, treatment effects were assessed following initial dose, the morning following nighttime dosing (to assess residual next day effects), and at steady state (i.e., following AM dosing on Day 3).
Time Frame: at time of peak concentration of drug (Tmax) on Day 1
Population: per protocol
Measure: Mean (Standard Deviation); unit: cm of deviation of lateral position
Groups:
- Tolperisone HCl 150 mg: 150 mg tolperisone tablets administered by mouth every 8 hours for 3 days
Arm/Group | Tolperisone HCl 150 mg | Placebo Oral Tablet | Cyclobenzaprine 10 mg Oral Tablet
Number analyzed (Participants) | 33 | 31 | 33
cm of deviation of lateral position | 29.3 (6.25) | 29.7 (6.37) | 38.6 (12.35)

2. Secondary Outcome: Standard Deviation of Lateral Position (SDLP) in Simulated Driving Test of Tolperisone Compared to Placebo on Day 2 Next Day Residual Effect
Description: SDLP measured by simulated driving performance of tolperisone compared to placebo on Day 2 prior to morning dosing to determine the next day residual effect or hangover of treatment
Time Frame: in the morning predose on Day 2 following nighttime dosing
Population: Per protocol population was analyzed per treatment group, therefore all subjects completing a treatment were included in the analysis
Measure: Mean (Standard Deviation); unit: cm of deviation from lateral position
Arm/Group | Tolperisone HCl 150 mg | Placebo Oral Tablet | Cyclobenzaprine 10 mg Oral Tablet
Number analyzed (Participants) | 33 | 31 | 33
cm of deviation from lateral position | 29.6 (7.08) | 29.9 (7.71) | 35.1 (10.37)

3. Secondary Outcome: Sleepiness Endpoint Karolinska Sleepiness Scale KSS
Description: assessment of self-reported motivation for driving performance where 1 equals alert and 9 equals extremely sleepy
Time Frame: at Tmax on Day 1
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolperisone HCl 150 mg | Placebo Oral Tablet | Cyclobenzaprine 10 mg Oral Tablet
Number analyzed (Participants) | 29 | 31 | 31
units on a scale | 3.3 (1.96) | 3.4 (1.99) | 5.6 (2.44)

4. Secondary Outcome: Steady State Standard Deviation of Lateral Position (SDLP) Day 3
Description: SDLP measured on Day 3 at steady state following 3 days of dosing three times per day to achieve steady state drug concentration and effect on outcomes
Time Frame: Day 3
Population: ITT
Measure: Mean (Standard Deviation); unit: cm deviation from lateral position
Arm/Group | Tolperisone HCl 150 mg | Placebo Oral Tablet | Cyclobenzaprine 10 mg Oral Tablet
Number analyzed (Participants) | 29 | 31 | 31
cm deviation from lateral position | 29.8 (6.68) | 29.6 (7.46) | 31.7 (7.9)

ADVERSE EVENTS:
Time Frame: The total duration of study participation was approximately 4 weeks including screening to follow up.
Description: No difference in definition.
Arm/Group | Tolperisone HCl 150 mg | Placebo Oral Tablet | Cyclobenzaprine 10 mg Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 15/33 | 12/31 | 20/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolperisone HCl 150 mg (N=33) | Placebo Oral Tablet (N=31) | Cyclobenzaprine 10 mg Oral Tablet (N=33)
dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) — dizziness
headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 5 (5) | 2 (2) | 10 (10) — sleepiness
dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
frequent bowel movement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
sluggishness (General disorders) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
skin exfoliation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
disturbance inattention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03353922/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03353922/SAP_001.pdf